CLINICAL TRIAL: NCT06046989
Title: BEAM: Building Emotional Awareness and Mental Health in Parenting. An App-based Intervention to Improve Parental Mental Health and Support Children's Brain Development.
Brief Title: Building Emotional Awareness and Mental Health in Parenting (BEAM)
Acronym: BEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital (Other); Provincial Health Services Authority British Columbia (Other); Brain Canada (Other); MindSea Development (Unknown); Workerbee.tv (Unknown)
Responsible Party: Principal Investigator, Lianne Tomfohr-Madsen, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB23-0759
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Parent Mental Health; Parenting; Child Mental Health; Child Development
Keywords: anxiety; depression; anger; brain imaging; parenting; behavioural neuroscience; child development; child mental health; eHealth
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: This study will include two arms and is a randomized controlled trial. For the experimental arm, a total of 120 participants will be enrolled in the BEAM group in cohorts of 24. The other 120 participants will be in the treatment-as-usual group where they will not have access to BEAM but will be able to access other resources or treatment.
Who Masked: Outcomes Assessor
Masking Description: Research assistants who are conducting the MRI brain imaging will be blinded to the participants' condition (i.e., whether they are in the control or experimental group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEAM Program (Experimental): The BEAM Program is delivered via mobile application, weekly check-ins, and peer coaching. BEAM includes videos with emotion-regulation strategies that come from the Unified Protocol (evidence-based treatment for depression and anxiety disorders) and Dialectical Behavior Therapy (DBT) to help with mental health, as well they focus on developing self-compassion and effective communication. There are also supportive parenting videos which focus on providing parents with emotion-focused parenting strategies, based on Tuning in to Kids® and Parent Management Training - The Oregon Model (PMTO), which aim to help parents better understand and respond to their child. There will be approximately 15-20 minutes of videos to watch weekly.
  Interventions: Behavioral: Building Emotion Awareness and Mental Health (BEAM)
- Treatment-As-Usual (No Intervention): This is the control arm of the study. It is designed to account for the potential effects of time on symptoms of depression, anxiety, and anger.

INTERVENTIONS:
Behavioral: Building Emotion Awareness and Mental Health (BEAM) — BEAM is based on best-practices in telehealth and science-based program design principles aimed at promoting parental mental health and supportive parenting. The BEAM Program mobile application is designed and managed by MindSea. The weekly one-on-one check-ins with peer coaches (parents who previously participated in another research group-based mental health intervention) will use the secure videoconferencing platform Zoom (Healthcare license) and direct messaging through the BEAM app. Peer coaches will also engage with participants on the community peer support forum. Monthly drop-in group peer support sessions will be facilitated by peer coaches and/or mental health professionals on the BEAM research team. The BEAM program's content emphasizes self-compassion, effective communication practices, and building social support networks.
  Arms: BEAM Program

SUMMARY:
Postpartum (child age 0-5 years) mental health problems are common, with prevalence rates ranging from 15-20% for depression, 3-43% for anxiety, and approximately 30% for anger. Depression, anxiety, and anger often occur comorbidly. If left untreated, these disorders can be long-lasting and lead to child behaviour problems, brain changes, and risk for later mental illness. We developed an app-based treatment for parental mental illness: Building Emotional Awareness and Mental Health in Parenting (BEAM). The BEAM program includes mental health and parenting videos, peer coaching, as well as a forum and drop-in Zoom sessions where parents can connect with each other to receive and provide social support. The program is supported by peer coaches (parents with lived experience of recovery from mental illness and who may have received emotion-focused parenting support) and supervised by clinically-trained staff. Peer coaches check-in with parents weekly to support their progress. Our study will see the BEAM app's effect on parent mental health, parenting stress, child behaviour, and child brain structure and function. 240 parents with high depression, anxiety, and/or anger symptoms will be recruited, with half forming the treatment-as-usual group.

DETAILED DESCRIPTION:
Although there are existing treatments for parental mental illness, there can be barriers to accessing care such as high cost and limited options in rural areas. This is troubling as untreated parental mental health symptoms can contribute to adverse consequences for both the parent and child. Thus, early intervention is critical to help prevent negative long-term effects. Digital resources can provide effective support, as they bypass many of the barriers associated with in-person interventions. The BEAM app was designed to combat these barriers and assist parents struggling with their mental health and the transition to parenthood. BEAM is a 12-week intervention with weekly videos about mental health and parenting for participants to watch. Exercises will be available so participants can practice new skills. Participants will also participate in weekly check-ins with peer coaches and have access to a secure forum where they can talk to other participants and receive social support. The BEAM Program also includes optional monthly drop-in sessions where parents can connect with each other in real time over Zoom.

Parent mental health (depression, anxiety, anger), parenting stress, and overreactive parenting will be assessed pre- and post-intervention, as well as 6 months post-intervention. Child behaviour and mental health will also be measured at all three timepoints (pre-, post-, and 6-months post-intervention). Child brain structure and function will be examined by MRI scans 6-months post-intervention. Participants will also receive brief wellness monitoring surveys in-app on a weekly basis.

There are three objectives for the present study:

1. Examine the effects of the BEAM program on parent mental health (including symptoms of depression, anxiety, and anger).
2. Examine the effects of the BEAM program on children's behaviour and mental health.
3. Examine the effects of the BEAM program on children's brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Parent is 18 years of age or older
* Must have a child who is 3-4 years old
* Must show clinically elevated symptoms of depression, anxiety, &/or anger
* Living in the Vancouver or Calgary area
* Parent is comfortable understanding, speaking, and reading English

Exclusion Criteria:

* Parent is under the age of 18
* Does not show clinically elevated symptoms of depression, anxiety, and/or anger
* History of attempted suicide or self-harm in the past 6 months
* Does not live in the Vancouver or Calgary area
* Child has serious genetic, neurological, or neurodevelopmental disorders that impact cognitive function or brain structure/function (e.g., Down Syndrome, epilepsy, etc.), or if they have contra-indications to MRI scanning (i.e., metal implants)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in parental mental health | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  Parent mental health will be a composite of symptoms of depression, anxiety, and anger. Depression symptoms will be measured via the 10-item Center for Epidemiologic Studies Depression Scale (CES-D; scores range from 0-30 with higher score indicating more severe symptoms). Clinically elevated depressive symptoms will be identified with a cut-off of >10. Anxiety symptoms will be measured via the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety short form (raw scores range from 7-35 with higher scores indicating more severe symptoms). Parent anger will be measured via PROMIS Anger (raw scores range from 5-25 with higher scores indicating more anger). T-score cut-offs of >60 will be used to identify those with clinically elevated anger and anxiety symptoms. An aggregate variable for parent mental health symptoms will be computed by converting scores on the CES-D, PROMIS Anxiety, and PROMIS Anger to standardized z-scores and then taking their average.

SECONDARY OUTCOMES:
Changes in parenting stress | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  The Parenting Stress Index (PSI) is a measure of parenting stress and interactional style. Scores range from 36-180; higher scores indicate greater parental stress.
Changes in parent self-efficacy | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  The Me as a Parent Scale- Short Form (MaaPs-SF) is a 4-item measure that will be used to examine parenting self-efficacy. Scores can range from 4-20, with higher scores indicating greater self-efficacy.
Changes in discipline practices | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  The Parenting Scale assesses the discipline practices of parents who have young children. The scores can range from 30-210; higher scores indicate more ineffective parenting discipline practices.
Changes in relationship satisfaction | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  The Couple Satisfaction Index assesses relationship satisfaction. Scores can range from 0-21; higher scores indicate greater relationship satisfaction.
Changes in household environment | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  The Chaos, Hubbub, and Order Scale will also be administered to capture the household environment. Scores can range from 0-15; higher scores indicate a more chaotic and disorganized environment.
Changes in children's behaviour | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  A parent will complete the Behaviour Assessment System for Children Third Edition (BASC-3) Parent Rating Scales-Preschool which assesses children's social-emotional functioning and behaviour. This is a 139-item questionnaire which provides T scores and percentile ranks. T scores have a mean of 50 and a standard deviation of 10.
Changes in children's mental health and development | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  This will be assessed using the Children's Somatic Symptoms Inventory-parent report (CSSI-8). The CSSI-8 scores can range from 0-32; higher scores indicate more somatic distress.
Children's structural brain connectivity | To be assessed 6 months post-intervention
  Children's structural brain connectivity will be assessed via MRI scans. A variety of images will be collected including anatomical (T1-weighted, T2-weighted) and diffusion-weighted MRI scans. Total scan duration is approximately 45 minutes. During the MRI scan, participants may watch a movie or video of their choice. The study team will work with participants to maximize their comfort during the scan, but children may choose to decline further time in the MRI scanner at any time. Following the MRI scan, images will be preprocessed and analyzed to identify key anatomical regions and the structural (i.e., white matter) connectivity between regions. Preprocessing and analysis will be conducted using popular neuroimaging tools including FSL, FreeSurfer, MRtrix, and R.
Children's functional brain connectivity | To be assessed 6 months post-intervention
  Children's functional brain connectivity will be assessed via MRI scans. A variety of images will be collected including anatomical (T1-weighted, T2-weighted), diffusion-weighted, and functional MRI scans. Total scan duration is approximately 45 minutes. During the MRI scan, participants may watch a movie or video of their choice. The study team will work with participants to maximize their comfort during the scan, but children may choose to decline further time in the MRI scanner at any time. Following the MRI scan, images will be preprocessed and analyzed to identify key anatomical regions and the functional (i.e., neuronal activity) connectivity between regions. Preprocessing and analysis will be conducted using popular neuroimaging tools including FSL, FreeSurfer, MRtrix, and R.
Children's phonological processing | To be assessed 6 months post-intervention
  Children's language ability will be partly assessed using the Phonological Processing subtest of the NEPSY second edition (NEPSY-II). Phonological Processing is a 22-item measure with scores ranging from 0-22, with higher scores indicating better word segment recognition. The subtest also has percentile rank scores based on normative data.
Children's speeded naming ability | To be assessed 6 months post-intervention
  Children's language ability will be partly assessed using the Speeded Naming subtest of the NEPSY-II. Speeded Naming is a 2-item measure with a maximum completion time of 300 seconds for naming 12 colours and 300 seconds for naming 12 shapes. A shorter completion time means more rapid access to and vocalization of names and shapes. The subtest also has percentile rank scores based on normative data.
Changes in parental sleep | To be assessed pre-intervention, immediately post-intervention, and 6-months post-intervention
  The PROMIS Sleep Disturbance- Short Form (PROMIS Sleep) will be used to assess parents' sleep. It is an 8-item measure with raw scores ranging from 8 to 40, where higher scores indicate greater sleep disturbance. Raw scores will be converted to T-scores which can be used to categorize sleep disturbance as "None to Slight," "Mild," "Moderate," or "Severe."
Adverse childhood experiences | To be assessed at pre-intervention
  The Adverse Childhood Experiences (ACEs) questionnaire will be administered to parents to examine what, if any, adverse experiences they had before the age of 18. It is an 11-item questionnaire that examines eight areas of adversity across three factors: Household Dysfunction (score range: 0-5), Physical/Emotional Abuse (score range: 3-9), Sexual Abuse (score range: 3-9).

CONTACTS AND LOCATIONS:
Overall Officials: Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of British Columbia; Catherine Lebel, PhD, Principal Investigator — University of Calgary; Leslie E Roos, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacKinnon AL, Simpson KM, Salisbury MR, Bobula J, Penner-Goeke L, Berard L, Rioux C, Giesbrecht GF, Giuliano R, Lebel C, Protudjer JLP, Reynolds K, Sauer-Zavala S, Soderstrom M, Tomfohr-Madsen LM, Roos LE. Building Emotional Awareness and Mental Health (BEAM): A Pilot Randomized Controlled Trial of an App-Based Program for Mothers of Toddlers. Front Psychiatry. 2022 Jun 24;13:880972. doi: 10.3389/fpsyt.2022.880972. eCollection 2022. PMID 35815022
- [Background] Xie EB, Simpson KM, Reynolds KA, Giuliano RJ, Protudjer JLP, Soderstrom M, Sauer-Zavala S, Giesbrecht GF, Lebel C, Mackinnon AL, Rioux C, Penner-Goeke L, Freeman M, Salisbury MR, Tomfohr-Madsen L, Roos LE. Building Emotional Awareness and Mental Health (BEAM): study protocol for a phase III randomized controlled trial of the BEAM app-based program for mothers of children 18-36 months. Trials. 2022 Sep 5;23(1):741. doi: 10.1186/s13063-022-06512-5. PMID 36064436